CLINICAL TRIAL: NCT03867409
Title: The United States Healthy Living Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB201801473 -N; 5R01CA207689-02 (NIH); OCR19177 (Other: UF OnCore)
Record Dates: First submitted 2019-03-01; First posted 2019-03-08 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study design will be a message design experiment for delivering a CRC intervention. Participants will receive a racially concordant virtual human message or a racially concordant text-based message based on their self-reported demographics (white or black).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Human (VH) Demographically Concordant - Black (Experimental): Participants received colorectal cancer screening information using a virtual human that matched their self-reported demographics.
  Interventions: Behavioral: message delivered via virtual technology
- Virtual Human (VH) Demographically Concordant - White (Experimental): Participants received colorectal cancer screening information using a virtual human that matched their self-reported demographics.
  Interventions: Behavioral: message delivered via virtual technology
- Text-Based Demographically Concordant - Black (Active Comparator): Participants received colorectal cancer screening information using a text-based message that matched their self-reported demographics.
  Interventions: Behavioral: message delivered via virtual technology
- Text-Based Demographically Concordant - White (Active Comparator): Participants received colorectal cancer screening information using a text-based message that matched their self-reported demographics.
  Interventions: Behavioral: message delivered via virtual technology

INTERVENTIONS:
Behavioral: message delivered via virtual technology — The intervention is precision messaging tailored to target audiences through development and evaluation of culturally sensitive, interactive messages about CRC screening delivered using VHT. The study will investigate whether interactive, tailored messages contribute to an overall enhancement of knowledge of CRC and screening options by eliciting positive attitudes and behaviors toward FIT screening.

SUMMARY:
The purpose of this study is to pilot test the efficacy of a patient-centered, tailored message intervention delivered via virtual human technology for increasing colorectal cancer (CRC) screening within guidelines. Although participation is not limited to these groups, the study team is particularly interested in the feasibility of the intervention for reaching racial/ethnic minority and rural patients.

DETAILED DESCRIPTION:
The primary goal of the study is to reduce colorectal cancer (CRC) morbidity and mortality by increasing CRC screening rates among the at-risk patient community and to reduce racial and geographic (rural vs. urban) disparities in CRC screening and mortality rates. To accomplish this long-term goal, this study aims to develop and test precision messaging tailored to target audiences through development and evaluation of culturally sensitive, interactive messages about CRC screening delivered using VHT. The study will investigate whether interactive, tailored messages contribute to an overall enhancement of knowledge of CRC and screening options by eliciting positive attitudes and behaviors toward FIT screening.

To date, there is no other study that has looked to partner specific message strategies and colorectal cancer screening with an emphasis on racial concordance and modality. As such, the researchers hope to shed new light on how, as health communicators, to more successfully engage target audiences to change attitudes and/or behaviors towards getting screened for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* reside within the United States but outside of Florida
* speak English
* are of either black or white racial background.
* are out-of-guidelines for colorectal cancer screening (>10 years for colonoscopy, >3 years for Cologuard, > 1 year for fecal immunochemical test)

Exclusion Criteria:

* does not meet the above criteria

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2105 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Krieger, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Human Demographically Concordant - Black: Participants receive colorectal cancer screening information using a virtual human that matches their self-reported demographics.
- Virtual Human Demographically Concordant - White: Participants received colorectal cancer screening information using a virtual human that matched their self-reported demographics.
Period: Overall Study
Arm/Group | Virtual Human Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human Demographically Concordant - White | Text-Based Demographically Concordant - White
Started | 333 | 330 | 722 | 720
Completed | 333 | 330 | 722 | 720
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White | Total
Number analyzed (Participants) | 333 | 330 | 722 | 720 | 2105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 290 | 295 | 549 | 508 | 1642
  >=65 years | 43 | 35 | 173 | 212 | 463
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 251 | 371 | 369 | 1237
  Male | 87 | 79 | 351 | 351 | 868
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 25 | 14 | 57
  Not Hispanic or Latino | 318 | 313 | 696 | 702 | 2029
  Unknown or Not Reported | 7 | 7 | 1 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 333 | 330 | 0 | 0 | 663
  White | 0 | 0 | 722 | 720 | 1442
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intention to Talk to Doctor About Colorectal Cancer Screening
Description: Measure: Intention to talk to doctor about colorectal cancer screening. Construct: Behavioral intention to communicate Item: The virtual appointment made me want to discuss colon cancer screening options with my doctor.
  Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate a lower intention to talk to a healthcare professional about colorectal cancer screening. Mean scores near 5 indicate a high intention to talk to a healthcare professional about colorectal cancer screening.
  No subscales
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.14 (1.13) | 4.0 (1.17) | 3.59 (1.26) | 3.48 (1.30)

2. Primary Outcome: Intention to Screen for Colorectal Cancer
Description: Measure: Intention to Screen for Colorectal Cancer Item: I want to get screened for colorectal cancer. Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate a lower intention to get screened for colorectal cancer. Mean scores near 5 indicate a higher intention to get screened for colorectal cancer.
  Construct: Behavioral intention to screen No subscales
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.03 (1.20) | 3.91 (1.21) | 3.57 (1.24) | 3.50 (1.28)

3. Primary Outcome: Intention to Talk About Screening With FIT
Description: Measure: Intention to Talk about Screening with FIT Item: I will talk to my healthcare provider about colon cancer screening with FIT.
  Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores closer to 1 indicate a lower intention to screen with FIT. Mean scores closer to 5 indicate a high intention to screen with FIT.
  Construct: Behavioral intention to screen with FIT No subscales
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.12 (1.16) | 4.03 (1.17) | 3.65 (1.27) | 3.50 (1.32)

4. Primary Outcome: Intention to Recommend Intervention (ALEX)
Description: Measure: Intention to Recommend Intervention (ALEX) Item: Imagine you received a link to ALEX from your healthcare provider. Would you like to share it by sending the link to someone? Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate a lower intention to recommend ALEX. Mean scores near 5 indicate a high intention to recommend ALEX.
  Construct: Behavioral intention to recommend ALEX No subscales
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 1.35 (0.48) | 1.36 (0.48) | 1.60 (0.49) | 1.66 (0.48)

5. Primary Outcome: Source Credibility
Description: Measure:
  Construct: Source Credibility
  Scale description: An 18-item unidimensional 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate that information provided by ALEX was perceived as not credible. Mean scores near 5 indicate the information provided by ALEX was perceived as highly credible. No subscales. The scale includes the following items:
  1. Intelligent-Unintelligent-Intelligent
  2. Untrained- Trained
  3. Doesn't care about me-Cares about me
  4. Dishonest- Honest
  5. Doesn't have my interests at heart-Has my interests at heart
  6. Untrustworthy-Trustworthy
  7. Inexpert -Expert
  8. Self-centered-Not self-centered
  9. Not concerned with me-Concerned with me
  10. Dishonorable-Honorable
  11. Uninformed-Informed
  12. Immoral-Moral
  13. Incompetent-Competent
  14. Unethical-Ethical
  15. Sensitive-Insensitive
  16. Stupid-Bright
  17. Phony-Genuine
  18. Not understanding-Understanding
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.54 (0.57) | 4.42 (0.64) | 4.35 (0.60) | 4.23 (0.64)

6. Primary Outcome: Argument Strength
Description: Construct: Argument Strength; Description: Argument Strength is a 9-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions of the strength of the argument about colon cancer screening. Mean scores near 1 indicate that ALEX's argument about colon cancer screening was perceived as not strong. Mean scores near 5 indicate that ALEX's argument about colon cancer screening was perceived as very strong. No subscales.
  1. The reason ALEX gives me for screening with FIT is believable
  2. The reason ALEX gives me for screening with FIT is convincing
  3. The reason ALEX gives me for screening with FIT is important to me
  4. ALEX helps me feel confident about how best to screen with FIT
  5. ALEX would help my friends screen with FIT
  6. ALEX encouraged me to screen with FIT
  7. ALEX encouraged me to avoid screening.
  8. I agree with ALEX's reasoning for screening
  9. ALEX gives a strong reason for screening with FIT
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.68 (0.62) | 4.57 (0.70) | 4.48 (0.75) | 4.39 (0.80)

7. Primary Outcome: Homophily
Description: Construct: Internal Homophily
  Scale: an 8-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions of their similarity to ALEX's characteristics. Mean scores near 1 indicate participants perceive strong dissimilarity to ALEX's characteristics. Mean scores near 5 indicate participants perceive strong similarity to ALEX's characteristics. No subscales. Items:
  1. Doesn't think like me-thinks like me
  2. Doesn't behave like me-Behaves like me
  3. Is different from me-Is similar to me
  4. Unlike me-Is like me
  5. Has a background different to mine-Has a background similar from mine
  6. Has morals unlike mine-Has morals like mine
  7. Looks different from me-Looks similar to me
  8. Is a different body size than I am-Has the same body size as I do
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.05 (1.18) | 3.04 (1.20) | 2.71 (1.16) | 2.75 (1.11)

8. Primary Outcome: Usability of App
Description: Construct: Usability of App; Description: Usability is a 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree). This scale measures participants' experience using the ALEX app. Mean scores near 1 indicate a negative experience using the ALEX app. Mean scores near 5 indicate a positive experience using the ALEX app. No subscales. Items:
  1. Enjoyable
  2. Easy to use
  3. Awkward
  4. Uncomfortable
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.48 (0.64) | 4.33 (0.78) | 4.30 (0.70) | 4.18 (0.72)

9. Primary Outcome: Perceived Severity
Description: Construct: Perceived Severity; Description: A 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions regarding the likelihood of developing colon cancer at some point in their lives. Mean scores near 1 indicate low severity, while mean scores near 5 indicate high severity. No subscales. Items:
  1. I am at risk for getting colon cancer in my lifetime.
  2. It is possible that I will get colon cancer in my lifetime.
  3. I am susceptible to getting colon cancer in my lifetime.
  4. It is likely that I will get colon cancer in my lifetime.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.47 (0.72) | 4.48 (0.68) | 4.55 (0.60) | 4.51 (0.62)

10. Primary Outcome: Perceived Susceptibility
Description: Construct: Perceived Susceptibility Description: Perceived Susceptibility is a 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) assessing participants' perceptions regarding being susceptible to developing colon cancer at some point in their lives. Mean scores near 1 indicate low susceptibility, while mean scores near 5 indicate high susceptibility. No subscales. Items:
  1. I am at risk for getting colon cancer in my lifetime.
  2. It is possible that I will get colon cancer in my lifetime.
  3. I am susceptible to getting colon cancer in my lifetime.
  4. It is likely that I will get colon cancer in my lifetime.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.10 (1.06) | 3.04 (1.06) | 3.35 (0.95) | 3.30 (0.95)

11. Primary Outcome: Response Efficacy
Description: Construct: Response Efficacy Description: A 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measured participants' perceptions of the effectiveness of FIT screening in detecting and preventing colon cancer. Mean scores near 1 indicate low perceived efficacy, while mean scores near 5 indicate high perceived efficacy. No subscales. Items:
  1. FIT screening leads to early detection if something is wrong.
  2. FIT screening leads to the detection of small abnormalities.
  3. FIT screening will help me find cancer early.
  4. FIT screening will decrease my chances of dying from colon cancer.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.09 (1.00) | 4.14 (0.92) | 4.16 (0.92) | 4.12 (0.90)

12. Primary Outcome: Self-Efficacy
Description: Construct: Self-Efficacy Description: A 12-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' confidence in completing FIT screening or a colonoscopy. Mean scores near 1 indicate low self-efficacy, while scores near 5 indicate high self-efficacy. No subscales. Items:
  1. I am confident that I can use the FIT
  2. Arranging my schedule to use the FIT is an easy thing to do
  3. FIT screening would be easy for me to do
  4. It would be easy for me to take a stool sample
  5. It would be easy for me to mail my kit back
  6. It would be easy for me to use all the tools in the kit
  7. I know how to collect a stool sample
  8. I am confident that I can get a colonoscopy
  9. Arranging my schedule to get a colonoscopy is an easy thing to do
  10. Finding time to get a colonoscopy would be difficult for me to do
  11. Screening for colon cancer with a colonoscopy would be easy for me to do
  12. It would be easy for me to get a colonoscopy
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.37 (0.73) | 4.32 (0.76) | 4.40 (0.69) | 4.27 (0.73)

13. Primary Outcome: Perceived Barriers
Description: Construct: Perceived Barriers Description: A 6-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) assessed participants' perceived obstacles to undergoing FIT screening. Mean scores closer to 1 indicate fewer perceived barriers. Mean scores closer to 5 indicate more perceived barriers. No subscales. Items:
  1. My doctor would never recommend the FIT.
  2. The FIT would be too expensive.
  3. The FIT would be too embarrassing.
  4. Preparation for the FIT is too hard.
  5. The FIT takes too much time.
  6. The FIT is difficult because it is too hard to understand all the instructions.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 1.86 (0.72) | 1.92 (0.70) | 1.95 (0.63) | 2.04 (0.68)

14. Primary Outcome: Perceived Benefits
Description: Construct: Perceived Benefits Description: A 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measured participants' perceptions of the benefits of FIT screening. Mean scores near 1 indicate low perceived benefits. Mean scores near 5 indicate high perceived benefits. No subscales. Items:
  1. The FIT will decrease my chances of dying from colon cancer.
  2. The FIT will help me not worry as much about colon cancer.
  3. I believe that if I had a normal screening test result, I wouldn't have to worry about developing colon cancer.
  4. I believe that when colon cancer is found early, it can be cured.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.2 (0.79) | 4.18 (0.75) | 4.18 (0.67) | 4.06 (0.72)

15. Primary Outcome: Comparative Risk Feedback
Description: Construct: Comparative Risk Feedback Description: A single-item unidimensional measure assessing participants' perceived risk of developing colon cancer compared to others on a 7-point Likert Scale. Mean scores near 1 indicate low perceived comparative risk. Mean scores near 7 indicate a high perceived risk of developing colon cancer compared to others. Item:
  1. Compared to the average person your age, gender, and race, how would you rate your chances of developing colon cancer in your life?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 5.18 (0.91) | 5.19 (1.01) | 5.15 (0.83) | 5.13 (0.81)

16. Primary Outcome: Cancer Information Overload
Description: Construct: Cancer Information Overload Description: A 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions regarding the amount and clarity of cancer-related information. Mean scores near 1 indicate lower overload. Mean scores near 5 indicate higher overload. No subscales. Items:
  1. There are so many different recommendations about preventing cancer, it's hard to know which ones to follow.
  2. There is not enough time to do all of the things recommended to prevent cancer.
  3. It has gotten to the point where I don't even care to hear new information about cancer.
  4. I feel overwhelmed by the amount of cancer information I am supposed to know.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 2.37 (0.94) | 2.49 (0.98) | 2.83 (0.91) | 2.97 (0.94)

17. Primary Outcome: Perceived Message Relevance
Description: Construct: Perceived Message Relevance Description: A 6-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions of how relevant and personalized the health message felt to them. Mean scores near 1 indicate low relevance. Mean scores near 5 indicate high relevance. No subscales. Items:
  1. The message seemed to be written personally for me.
  2. The message was very relevant to my situation.
  3. The message was applicable to me.
  4. The message was very customized to me.
  5. This message was manipulative.
  6. This message was misleading.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.75 (1.12) | 3.66 (1.15) | 3.60 (1.05) | 3.48 (1.0)

18. Primary Outcome: Trust in Physician
Description: Construct: Trust in Physician Description: An 11-item 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring physician trust. Mean scores near 1 indicate low trust, while scores near 5 indicate high trust. No subscales. Items:
  1. I doubt that my doctor really cares about me as a person
  2. My doctor usually puts my needs first
  3. I trust my doctor so much I always try to follow his/her advice
  4. If my doctor tells me something is so, then it must be true
  5. I sometimes distrust my doctor's opinion
  6. I trust my doctor's judgments about my medical care
  7. I feel my doctor does not do everything he/she should about my medical care
  8. I trust my doctor to put my medical needs above all other considerations
  9. My doctor is well qualified to manage my medical problems
  10. I trust my doctor to tell me if a mistake was made about my treatment
  11. I sometimes worry that my doctor may not keep the information we discuss totally private
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.86 (1.08) | 3.86 (1.03) | 3.66 (1.06) | 3.65 (1.02)

19. Primary Outcome: Patient-Provider Communication
Description: Construct: Patient-Provider Communication Description: A 5-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' perceptions of how well their doctor communicates with them. Mean scores near 1 indicate poor communication. Mean scores near 5 indicate good communication. No subscales. Items:
  1. I receive enough understandable information from my doctor/healthcare provider to make good decisions about my health.
  2. I feel rushed during visits.
  3. My doctor/healthcare provider involves me in decisions about my health care treatment.
  4. I feel uncomfortable asking my doctor for tests or information if he/she doesn't mention it.
  5. My doctor/healthcare provider understands my health needs.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 4.13 (0.99) | 4.05 (0.96) | 3.86 (1.05) | 3.88 (0.94)

20. Primary Outcome: Patient General Health
Description: Construct: Patient General Health Description: A 3-item unidimensional measure assessing participants' overall health and pain levels on 5-point Likert Scales. Mean scores near 1 indicate low general health. Mean scores near 5 indicate high general health. Items:
  1. In general, would you say your health is: (1=Poor, 5=Excellent)
  2. How much bodily pain have you had during the past 4 weeks? (1= Very severe, 5= None)
  3. During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? (1 = Extremely, 5= Not at all)
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.09 (0.87) | 3.18 (0.93) | 3.20 (0.93) | 3.17 (0.95)

21. Primary Outcome: Health Literacy (eHeals)
Description: Construct: Health Literacy (eHeals) Description: An 8-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) measuring participants' confidence in using the internet for health-related information. Mean scores near 1 indicate low health literacy. Mean scores near 5 indicate high health literacy. No subscales. Items:
  1. I know how to find helpful health resources on the Internet.
  2. I know how to use the Internet to answer my health questions.
  3. I know what health resources are available on the Internet.
  4. I know where to find helpful health resources on the Internet.
  5. I know how to use the health information I find on the Internet to help me.
  6. I have the skills I need to evaluate the health resources I find on the Internet.
  7. I can tell high quality from low quality health resources on the Internet.
  8. I feel confident in using information from the Internet to make health decisions.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.98 (0.90) | 4.02 (0.90) | 3.83 (0.88) | 3.75 (0.93)

22. Primary Outcome: Interpersonal Distance
Description: Construct: Interpersonal Distance Description: A 4-item unidimensional 5-point Likert scale (1=strongly disagree/5=strongly agree) that measures participants' perceptions of the virtual human's presence. Mean scores near 1 indicate low perceived presence. Mean scores near 5 indicate high perceived presence. No subscales. Items:
  1. I perceive that I am in the presence of Alex in the room with me.
  2. I feel that Alex is aware of my presence.
  3. The thought that Alex is not a real person crosses my mind often.
  4. I perceive Alex as being only a computerized image, not as a real person.
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.49 (0.83) | 3.39 (0.88) | 3.37 (0.82) | 3.26 (0.82)

23. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Sad
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Sad
  Description: We measured participant's emotional attitudes of sadness towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of sadness regarding FIT screening. Mean scores near 5 indicate strong feelings of sadness regarding FIT screening. Item:
  1. How much sadness would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 1.59 (0.92) | 1.72 (1.11) | 1.67 (0.97) | 1.72 (1.0)

24. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Worried
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Worried
  Description: We measured participant's emotional attitudes of worry towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of worry regarding FIT screening. Mean scores near 5 indicate strong feelings of worry regarding FIT screening. Item:
  1. How much worried would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 2.31 (1.3) | 2.51 (1.37) | 2.4 (1.26) | 2.47 (1.31)

25. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Relieved
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Relieved Description: We measured participant's emotional attitudes of relief towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of relief regarding FIT screening. Mean scores near 5 indicate strong feelings of relief regarding FIT screening. Item:
  1. How relieved would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.53 (1.28) | 3.36 (1.34) | 3.28 (1.27) | 3.05 (1.28)

26. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Tense
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Tense
  Description: We measured participant's emotional attitudes of tensity towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of tenseness regarding FIT screening. Mean scores near 5 indicate strong feelings of tenseness regarding FIT screening. Item:
  1. How tense would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 2.50 (1.33) | 2.71 (1.41) | 2.51 (1.31) | 2.63 (1.34)

27. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Anxious
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Anxious
  Description: We measured participant's emotional attitudes of anxiety towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of anxiousness regarding FIT screening. Mean scores near 5 indicate strong feelings of anxiousness regarding FIT screening. Item:
  1. How anxious would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 2.58 (1.37) | 2.82 (1.41) | 2.64 (1.30) | 2.76 (1.36)

28. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Calm
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Calm
  Description: We measured participant's emotional attitudes of calmness towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of calmness regarding FIT screening. Mean scores near 5 indicate strong feelings of calmness regarding FIT screening. Item:
  1. How calm would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 3.30 (1.30) | 3.18 (1.37) | 3.09 (1.26) | 3.00 (1.31)

29. Primary Outcome: Attitudes Towards Fecal Immunochemical Test (FIT) - Afraid
Description: Construct: Attitudes towards Fecal Immunochemical Test (FIT) - Afraid
  Description: We measured participant's emotional attitudes of fear towards FIT using single-items on a 5-point Likert scale (1=not at all, 5=very much). Mean scores near 1 indicate little to no feelings of fear regarding FIT screening. Mean scores near 5 indicate strong feelings of fear regarding FIT screening. Item:
  1. How afraid would you feel if a doctor asked you to get screened for colon cancer using FIT?
Time Frame: immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
Number analyzed (Participants) | 333 | 330 | 722 | 720
units on a scale | 2.28 (1.31) | 2.48 (1.37) | 2.32 (1.25) | 2.40 (1.29)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 months.
Description: During the study, 2,105 participants were monitored/assessed for other (non-serious) adverse events, but none were observed.
Arm/Group | Virtual Human (VH) Demographically Concordant - Black | Text-Based Demographically Concordant - Black | Virtual Human (VH) Demographically Concordant - White | Text-Based Demographically Concordant - White
All-Cause Mortality (participants affected / at risk) | 0/333 | 0/330 | 0/722 | 0/720
Serious Adverse Events (participants affected / at risk) | 0/333 | 0/330 | 0/722 | 0/720
Other Adverse Events (participants affected / at risk) | 0/333 | 0/330 | 0/722 | 0/720

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03867409/Prot_SAP_ICF_000.pdf